CLINICAL TRIAL: NCT05614310
Title: Early Detection Of Alzheimer's Disease With GlucoCEST MRI: A Feasibility Study.
Brief Title: Detecting Early Alzheimer's Using MR
Acronym: DREAMER
Status: Recruiting | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-001-22; TCS/21/03 (Other Grant/Funding Number: Chief Scientist Office); 22\LO\0347 (Other: National Health Service Research Ethics Committees); 308185 (Other: IRAS (Integrated Research Application System))
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Alzheimer Disease
Keywords: Magnetic Resonance Imaging (MRI); Glucose Chemical Exchange Saturation Transfer (CEST)
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy; Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Development Group 1 (N = 10) (Development Phase): Development group participants (N = 10) will undergo 1 magnetic resonance imaging (MRI) sessions. Before and after their MRI scan participants will be given a pinprick blood sugar test.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Other: Blood Glucose Assessment
- Patients (N = 20) (Clinical Phase): Patients (N = 20) will attend 2 visits up to 1 week apart. Patients will be asked to have a no-sugar diet and take no exercise for 24 hours before each visit and to avoid eating 6 hours before scan.
  Visit 1: Patients will undergo a positron emission tomography (PET) assessment. Before and after their PET assessment patients will be given a pinprick blood sugar test. PET assessment:
  Visit 2: Patients will undergo MRI assessment. Before and after their MRI scan patients will be given a pinprick blood sugar test. Healthy controls will complete cognitive assessments.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Other: Blood Glucose Assessment; Other: Positron Emission Tomography (PET); Other: Cognitive Assessment
- Healthy Controls (N = 20) (Clinical Phase): Healthy controls (N = 20) will attend 2 visits up to 1 week apart. Healthy controls will be age matched (+/- 3 years) and sex matched to the patient group. Healthy controls will be asked to have a no-sugar diet and take no exercise for 24 hours before each visit and to avoid eating 6 hours before scan.
  Visit 1: Healthy Controls will undergo a positron emission tomography (PET) assessment. Before and after their PET assessment patients will be given a pinprick blood sugar test. PET assessment:
  Visit 2: Healthy Controls will undergo MRI assessment. Before and after their MRI scan patients will be given a pinprick blood sugar test. Healthy controls will complete cognitive assessments.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Other: Blood Glucose Assessment; Other: Positron Emission Tomography (PET); Other: Cognitive Assessment
- Development Group 2 (N = 10) (Development Phase): To investigate the repeatability of MRI assessment, 10 development phase healthy volunteers will be recruited to undergo two repeated study assessments. The second visit will be between 7 and 14 days after their first visit. The second repeated study assessment will follow the same procedure as the first visit, consisting of blood glucose assessment and MRI assessment. Participants will be advised to fast from mid-night and avoid eating breakfast.
  Interventions: Other: Magnetic Resonance Imaging (MRI); Other: Blood Glucose Assessment

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — Participants will be asked to lie in the MRI scanner while we collect 3D T1- and T2-weighted images and a 3D FLAIR image to exclude pathology (e.g. stroke). Participants will ingest a glucose solution (75 g Dextrose) so dynamic glucoCEST images can be acquired to measure glucose uptake and clearance.
Other: Blood Glucose Assessment — A blood testing meter will be used to measure the blood sugar levels before and after the scans. Normal reading for a nondiabetic person after fasting is 70-99 mg/dl (3.9-6 mmol/L). If abnormal blood sugar levels are detected (sugar levels outside the above normal range), the participant will no longer be eligible for the study and they will be withdrawn.
Other: Positron Emission Tomography (PET) — Participants will be administered a radioactive glucose analogue, 2-deoxy-2-(18F) fluoro-D-glucose (18FDG) through a canula inserted into a vein in the arm or hand and asked to sit quietly for 1 h. After 1 h they will be asked to lie quietly and without talking in the PET scanner and a PET brain scan will be performed.
  Groups: Healthy Controls (N = 20) (Clinical Phase); Patients (N = 20) (Clinical Phase)
Other: Cognitive Assessment — Participants will be asked to undertake two cognitive tests (the Alzheimer's Disease Assessment Scale ADAS-cog test and the Mini Mental State Examination test - MMSE). These are standard clinical tests used to determine cognitive dysfunction in Alzheimer's disease.
  Groups: Healthy Controls (N = 20) (Clinical Phase); Patients (N = 20) (Clinical Phase)

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia, affecting approximately 10% of individuals aged ≥ 65. Most available treatments aim at controlling symptoms at an early stage rather than providing a cure. Therefore, an accurate and early diagnosis of AD with appropriate management will slow the progression of the condition. Reduced cerebral glucose levels have been observed in patients with early AD. Glucose hypometabolism can be assessed by administering a radioactive glucose analogue, 2-deoxy-2-(18F) fluoro-D-glucose (18FDG), and imaging with PET (positron emission tomography). The high cost and limited availability of PET-CT (PET - computed tomography) still hamper its general clinical application. Moreover, the use of radioactive tracers in combination with the additional ionizing radiation of CT is not suitable for repeated measurements. Therefore, currently, the provisional diagnosis of AD is still based on the combination of clinical history, neurological examination, cognitive testing over a period of time, and structural neuroimaging. This has major time and resource implications.

A radically different and highly innovative means for imaging glucose with magnetic resonance imaging (MRI) has now been established, exploiting the interaction between hydroxyl protons in glucose and the protons in water; the method is termed glucose Chemical Exchange Saturation Transfer (glucoCEST). GlucoCEST MRI is a method that has no reliance on radiolabelled glucose analogues and could become widely implemented in clinic practice. We therefore aim to investigate the potential of glucoCEST MRI in Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common cause of dementia, affecting approximately 10% of individuals aged ≥ 65. Most available treatments aim at controlling symptoms at an early stage rather than providing a cure. Therefore, an accurate and early diagnosis of AD with appropriate management will slow the progression of the condition. Reduced cerebral glucose levels have been observed in patients with early AD. Glucose hypometabolism can be assessed by administering a radioactive glucose analogue, 2-deoxy-2-(18F) fluoro-D-glucose (18FDG), and imaging with PET (positron emission tomography). The high cost and limited availability of PET-CT (PET - computed tomography) still hamper its general clinical application. Moreover, the use of radioactive tracers in combination with the additional ionizing radiation of CT is not suitable for repeated measurements. Therefore, currently, the provisional diagnosis of AD is still based on the combination of clinical history, neurological examination, cognitive testing over a period of time, and structural neuroimaging. This has major time and resource implications.

A radically different and highly innovative means for imaging glucose with magnetic resonance imaging (MRI) has now been established, exploiting the interaction between hydroxyl protons in glucose and the protons in water; the method is termed glucose Chemical Exchange Saturation Transfer (glucoCEST). GlucoCEST MRI is a method that has no reliance on radiolabelled glucose analogues and could become widely implemented in clinic practice. We believe that glucoCEST MRI has the potential to replace FDG-PET and improve patient healthcare as part of a routine clinical pathway in very early detection of AD.

The study will include 20 healthy volunteers for developing glucoCEST in the clinical 3T MRI scanner (development phase) and 20 volunteers without AD and 20 patients with clinically diagnosed AD (clinical phase). All participants will have a 3T brain MRI scan after they receive oral glucose. The participants in the clinical phase will have a 3T brain MRI scan, a brain PET scan and they will also undertake two cognitive tests.

The glucose uptake and clearance rate in the brain will be measured from PET and MRI scans and compared between groups and imaging modalities. Sensitivity and specificity of glucoCEST to detect AD will be also calculated.

Primary Objective: To estimate the sensitivity of glucose uptake as measured by glucoCEST MRI in patients with AD compared with age and sex matched controls.

Secondary objective: To investigate if the glucose uptake as measured by glucoCEST MRI is related to the glucose uptake as measured in FDG-PET.

The main aims of the study are:

1. To determine normal uptake and clearance rates of glucose in the brain as measured by dynamic glucoCEST MRI at 3T
2. To compare glucose uptake as measured by glucoCEST MRI and FDG-PET.
3. To compare glucose uptake as measured by glucoCEST MRI in patients with AD and age and sex matched controls.

ELIGIBILITY:
Inclusion Criteria:

Development phase:

Controls (development group) must:

* be > 18 years
* consent to the study
* not report problems with memory.

Clinical phase

Patients must:

* be ≥ 65 years,
* able to provide informed consent to the study
* have been clinically diagnosed with AD by the mental health team.

Controls must:

* be ≥ 65 years
* able to provide consent to the study
* have a normal score in the ADAS-cog test and the Mini Mental State Examination test (MMSE)
* not report problems with memory.

Exclusion Criteria:

Subjects will not be considered if they:

* have a history of diabetes,
* have history of a major stroke (mini-stroke/Transient Ischaemic Attacks or lacunar stroke are acceptable),
* have contra-indications to MRI scanning such as implantable cardiac devices
* have family history in AD, to exclude possible gene mutations associated with AD
* have advanced AD who lack the capacity to consent.
* Are pregnant (for developmental phase)
* are unable to read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Target population: For the methods development phase, 20 healthy volunteers (age 18 years and above) without contra-indications to MRI will be recruited. Twenty patients with clinically diagnosed AD and 20 age-matched controls (+/- 3 years) will be recruited to test the clinical feasibility of glucoCEST.
  As a feasibility study, the current work is unlikely to cover the full representative range of AD patients with diverse phenotypes. Its key purpose is to explore whether the proposed technique will show different glucose uptake between those with normal cognition and those with early AD. Further the purpose of future clinical use will be to detect AD in its early stage where clinical manifestations of AD are either subclinical or very mild. We will ensure that the sample is representative of the age range of AD patients, as well as sex balanced.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PET glucose measurement | 2 years
  Dynamic frames from FDG-PET will be summed and normalised to the cerebellum using MATLAB (MathWorks Inc., USA). Standardised uptake values (SUVs) from PET will then be calculated. Regions of interests (ROIs) will derived from normalisation to the standard Desikan Killiany atlas. Average SUV from PET will be calculated from each ROI in MATLAB.
  Glucose uptake (maximum ΔS/So) with units of ratio.
  Clearance (rate of decrease of ΔS/So) values with units of ratio.
CEST-MRI glucose measurement | 2 years
  Dynamic frames from CEST MRI will be summed and normalised to the cerebellum using MATLAB (MathWorks Inc., USA). Standardised uptake values (SUVs) will be calculated in regions of interests (ROIs) derived from normalisation to the standard Desikan Killiany atlas. Average SUV from each ROI, the glucose uptake (maximum ΔS/So) and clearance (rate of decrease of ΔS/So) values from patients and controls will be calculated using MATLAB.
  Glucose uptake (maximum ΔS/So) with units of ratio.
  Clearance (rate of decrease of ΔS/So) values with units of ratio
Sensitivity and specificity of CEST-MRI glucose measurements | 2 years
  A neuroradiologist blinded to the diagnosis of each participant will be asked to report the scans in a similar way to an FDG-PET scan. Sensitivity and specificity of glucoCEST to detect AD by estimating the proportion of true positives and true negatives respectively will be determined. To demonstrate the feasibility of glucoCEST in differentiating AD patients from controls, group comparisons of glucose (paired samples t-tests as implemented by SPSS) uptake values between patients and controls and of glucose clearance values between patients and controls will be performed.
  Sensitivity and specificity values with units of ratio.
Repeatability of CEST-MRI glucose measurement | 2 years
  To investigate the repeatability of MRI assessment, 10 out of 20 development phase healthy volunteers will be recruited to undergo a second repeated study assessment visit between 7 and 14 days after their first visit.
  Coefficient of variation values with units of percent.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Waiter, PhD, Study Chair — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kukull WA, Higdon R, Bowen JD, McCormick WC, Teri L, Schellenberg GD, van Belle G, Jolley L, Larson EB. Dementia and Alzheimer disease incidence: a prospective cohort study. Arch Neurol. 2002 Nov;59(11):1737-46. doi: 10.1001/archneur.59.11.1737. PMID 12433261
- [Background] Bloudek LM, Spackman DE, Blankenburg M, Sullivan SD. Review and meta-analysis of biomarkers and diagnostic imaging in Alzheimer's disease. J Alzheimers Dis. 2011;26(4):627-45. doi: 10.3233/JAD-2011-110458. PMID 21694448
- [Background] Marcus C, Mena E, Subramaniam RM. Brain PET in the diagnosis of Alzheimer's disease. Clin Nucl Med. 2014 Oct;39(10):e413-22; quiz e423-6. doi: 10.1097/RLU.0000000000000547. PMID 25199063
- [Background] Tolomeo D, Micotti E, Serra SC, Chappell M, Snellman A, Forloni G. Chemical exchange saturation transfer MRI shows low cerebral 2-deoxy-D-glucose uptake in a model of Alzheimer's Disease. Sci Rep. 2018 Jun 22;8(1):9576. doi: 10.1038/s41598-018-27839-7. PMID 29934551
- [Background] Wang J, Weygand J, Hwang KP, Mohamed AS, Ding Y, Fuller CD, Lai SY, Frank SJ, Zhou J. Magnetic Resonance Imaging of Glucose Uptake and Metabolism in Patients with Head and Neck Cancer. Sci Rep. 2016 Jul 27;6:30618. doi: 10.1038/srep30618. PMID 27461165
- [Background] Kim M, Torrealdea F, Adeleke S, Rega M, Evans V, Beeston T, Soteriou K, Thust S, Kujawa A, Okuchi S, Isaac E, Piga W, Lambert JR, Afaq A, Demetriou E, Choudhary P, Cheung KK, Naik S, Atkinson D, Punwani S, Golay X. Challenges in glucoCEST MR body imaging at 3 Tesla. Quant Imaging Med Surg. 2019 Oct;9(10):1628-1640. doi: 10.21037/qims.2019.10.05. PMID 31728307